CLINICAL TRIAL: NCT01994798
Title: Prospective, Non-randomized, Multicentre, Observational Registry to Assess Clinically Relevant Benefit of Performing the Whole PTA Procedure Using the Rapid Exchange (RX) Devices.
Brief Title: Rapid Exchange Devices Observational Registry.
Acronym: RXRegistry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T122E2
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Peripheral (Lowr Extremity) Arterial Disease.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This registry is designed to assess the clinically relevant benefits of balloon angioplasty and stenting in superficial femoral and popliteal artery, using rapid exchange technology.

DETAILED DESCRIPTION:
This registry is designed to assess the clinically relevant benefits of balloon angioplasty and stenting in superficial femoral and popliteal artery, using rapid exchange technology

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic one or two legs ischemia, requiring treatment of SFA or popliteal artery
* Rutherford classification 2-5
* Single lesion with recoiling/dissection/restenosis after balloon angioplasty or de novo lesions with stenosis or occlusion,
* Target vessel reference diameter ≥4mm and ≤7mm (by visual estimate)
* At least one patent (less than 50% stenosis) tibioperoneal run-off vessel confirmed by baseline angiography
* Patient is suitable candidate for femoral-popliteal artery bypass surgery

Exclusion Criteria:

* Female of child-bearing potential.
* Previous bypass surgery
* In stent restenosis as a target lesion
* Scheduled staged procedure of multiple lesions within the ipsilateral iliac or popliteal arteries within 30 days after index procedure.
* Co-existing aneurysmal disease of the abdominal aorta, iliac or popliteal arteries
* Acute thrombophlebitis or deep venous thrombosis
* Hemodynamic instability
* Untreated inflow disease of the ipsilateral pelvic arteries (more than 50 percent stenosis or occlusion),
* Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy
* Known intolerance to study medications, contrast agents or nitinol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with one lesion located in Superficial Femoral Artery(SFA) or popliteal artery planned to be treated as per hospital practice with plain old balloon angioplasty and nitinol stent using monorail (rapid exchange) delivery system.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Safety: composite of all-cause death, amputation, TVR, stroke or bleeding (BARC ≥ 3) up to 1 month | From start up to 30 Days post procedure.
Total contrast media volume given during the procedure. | During procedure

SECONDARY OUTCOMES:
Total duration of the procedure | During procedure
Total fluoroscopy time | During procedure
Total radiation dose given | During procedure
Technical success defined as a successful access and balloon angioplasty followed by stent placement with achieved recanalization determined by less than 30% residual stenosis by angiography at the baseline procedure. | Pre- and post-procedure
Clinical success defined as technically successful procedure without the events considered in safety composite endpoint (all-cause death, amputation, TVR, stroke or bleeding (BARC ≥ 3) up to 1 month. | During procedure
Total acute complication rate defined as any device- or procedure- related complication up to 1 month post procedure. | Up to 30 Days post procedure
Total acute device related complication rate defined as any device complication up to 1 month post procedure. | Up to 30 Days post procedure
Ankle-Brachial Index (ABI) improvement at 30 days. | 30 Days post procedure
Improvement of the Rutherford index at 30 days. | 30Days post procedure
Walking distance at 30 days compared with walking distance before procedure. | 30 Days post procedure
Bleeding complication as per BARC definitions. | Up to 30 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Martinez, Principal Investigator — Centre Hospitalier Universitaire (CHU) Liège; Omar Andrés Navarro, Principal Investigator — Hospital Universitari Dr. Josep Trueta de Girona; Josua Van den Berg, Principal Investigator — Ospedale Regionale di Lugano
Locations (9):
- Belgium (5):
  - Onze-Lieve-Vrouwziekenhuis (OLV) Aalst, Aalst
  - GasthuisZusters Antwerpen (GZA) Ziekenhuizen, Antwerp
  - Centre Hospitalier Régional (CHR) du Val de Sambre, Auvelais-Val de Sambre
  - Jessa Ziekenhuis, Hasselt
  - Centre Hospitalier Universitaire (CHU) Liège, Liège
- Spain (4):
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitari Dr. Josep Trueta de Girona, Girona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Valladolid, Valladolid